CLINICAL TRIAL: NCT05681286
Title: C-reactive Protein to Serum Albumin Ratio in Type 2diabetic Patients With Diabetic Nephropathy
Brief Title: CRP to Serum Albumin Ratio in Type 2 DM é Diabetic Nephropathy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Shymaa shahhat Abodahab, Investigator, Assiut University
Other Study IDs: CAR level in type 2 DM
Record Dates: First submitted 2022-12-25; First posted 2023-01-12 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2022-12

CONDITIONS: Type 2 DM /Diabetic Nephropathy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
we aimed to compare C-reactive protein to serum albumin ( CAR) level of the T2DM patients with DN to those T2DM without DN

DETAILED DESCRIPTION:
Diabetic Nephropathy (DN) is a serious complication of Diabetes Mellitus associated with chronic and low-grade inflammatory burden affects around 30 % of diabetic patients It is the leading cause of end-stage renal failure worldwide and associated with cardio vascular diseases and increases mortality of diabetic patients It characterized by persistent albuminuria, raise in arterial blood pressure ,decrease in glomerular filtration rate (GFR) It associated with chronic low grade inflammation that's leads to increase glucose and activities inflammation Despite of the pathogenesis of DN is multifactorial, but local inflammatory process may result from both the metabolic and hemodynamic affection seen in DN sustained diabetes-related metabolic and haemodynamic perturbations can induce subclinical low-grade renal inflammation and drive kidney from repair response to damage process, eventually to renal fibrosis Chronic inflammatory processes not only play a principle role in the progression of micro vascular but also macro vascular complications in type 2 diabetes mellitus. An association between low -grade inflammation and type 2 diabetes has been described in recent studies .C- reactive protein to serum albumin ratio has attracted great attention recently , and used as biomarker in detection disease severity

, since type 2 Diabetes Mellitus and Diabetic Nephropathy(DN) is associated with low grade inflammation in recent studies. In this study investigator presume that C-reactive protein to serum albumin ratio ( CAR )levels could be associated with the progression of DN in patients with T2DM.

ELIGIBILITY:
Inclusion Criteria All type 2diabetic patients

Exclusion Criteria:

* Type 1 diabetes is , patient t with liver cirrhosis, patient with active infection ,pregnant women,patients with cancer

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: type 2 DM patients
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2023-08-04 (Estimated); Primary Completion 2024-08-04 (Estimated); Study Completion 2025-08-04 (Estimated)

PRIMARY OUTCOMES:
C-reactive protein to serum albumin ratio in type 2diabetic patients with diabetic nephropathy | Baseline
  comparison between CAR level è type 2 diabetic nephropathy patient and those without nephropathy

CONTACTS AND LOCATIONS:
Overall Officials: Salah Argoon, Study Chair — Assuit u; Alshaimaa sayed, Study Chair — Assiut University